CLINICAL TRIAL: NCT04164264
Title: Genetic Differences in Pharmacodynamic Safety Endpoints With Propofol Anaesthesia in Children
Brief Title: Genetic Differences in Propofol Pharmacodynamics in Children
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University of British Columbia (Other)
Collaborators: BC Children's Hospital Research Institute (Other)
Responsible Party: Principal Investigator, Simon Whyte, Staff Anesthesiologist, University of British Columbia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: H19-00188
Record Dates: First submitted 2019-11-06; First posted 2019-11-15 (Actual); Last update posted 2024-04-22 (Actual); Status verified 2024-04

CONDITIONS: Anesthesia
Keywords: Propofol
MeSH Terms: interventions — Propofol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Intravenous Propofol Infusion (Experimental): Quantification of the dose of propofol required to produce loss of consciousness and apnea.
  Interventions: Drug: Propofol

INTERVENTIONS:
Drug: Propofol — At T0, a propofol infusion at a rate of 1.5 mg/kg/min will be started until apnea is achieved. Loss of consciousness will be defined clinically using loss of eyelash reflex (TLOER) and tolerance of nasal cannulae (TNC), tested every 10 sec., and by a BIS <60 for 30 sec. (TBIS). Apnea will be defined as absence of end-tidal CO2 for at least 20 seconds (TAPNEA). A saliva sample with be taken under anesthesia for genome-wide association study and principal component analysis.
  Other Names: Propofol Injection 1%

SUMMARY:
Propofol is an extensively utilized intravenous sedative and general anesthetic. However, propofol has a narrow therapeutic index, and this means that there is only a small difference in the dose required to produce loss of consciousness and the dose required to produce potentially life-threatening effects such as loss of protective airway reflexes and cessation of spontaneous breathing. Moreover, there is substantial variation between individuals in the doses required to achieve these pharmacodynamic endpoints.

Given the inexorable rise in demand for pediatric sedation and the increasing use of propofol in sedation protocols by non-anaesthesiologists, the purpose of this study is to refine the propofol dosing recommendations to account for pharmacogenomic variability to make procedural sedation safer for children. Experienced users already adjust for age and body weight. This study may enable further refinements according to sex and - novelly - ancestry.

DETAILED DESCRIPTION:
Hypothesis:

The investigators hypothesize that examination of genome-wide association study (GWAS) findings will enable the investigators to provide pharmacogenomic insights into clinically observed - and, with this study, quantified - differences in propofol requirements for loss of consciousness (LOC) and apnea in children. It is further hypothesized that the distribution of allelic variants in these pharmacogenes may differ between children of different genomic ancestry.

Objectives:

Primary: (i) To describe and quantify doses of propofol required to produce loss of consciousness and apnea in children of differing ages, sex and self-identified countries of origin. (ii) To identify genomic associations that may explain variability, and generate hypotheses for further study. (iii) To identify genomic ancestry and examine how pharmacogene allele variants that may explain the findings of (i) above are distributed across genomic ancestries.

Secondary: To examine the correlation between self-identified countries of family origin and genomic ancestry.

Methods:

Prospective, non-randomized, single cohort study of two pharmacodynamic endpoints (loss of consciousness and apnea), in children requiring propofol anesthesia, with subsequent genome-wide association study (GWAS) and principal component analysis (PCA) to examine, respectively, pharmacogenomic explanations for pharmacodynamic variability and genomic ancestry.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 3 to ≤ 18
* ASA physical status classification I-III
* Intravenous induction resulting in apnea clinically appropriate and indicated

Exclusion Criteria:

* Age < 3 or >18
* ASA physical status IV-V
* Propofol induction to apnea not indicated or feasible
* Sedative premedication
* Severe neurological impairment, expected to reduce propofol requirement as judged by the clinical experience of the anaesthetist
* Weight <3%ile or >97%ile for age

Ages: 3 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 360 (Actual)
Dates: Start 2020-03-11 (Actual); Primary Completion 2023-10-26 (Actual); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Dose of propofol required to produce loss of consciousness | Loss of consciousness will be expected to occur somewhere between 120-180 seconds after commencing the induction infusion.
  Loss of consciousness will be defined clinically when there is a loss of eyelash reflex, a tolerance of nasal cannulae, and when the Bispectral Index <60 for 30 sec.
Dose of propofol required to produce apnea | Apnea will be expected to occur within 10 min after commencing the induction infusion.
  Apnea will be defined as absence of end-tidal CO2 for at least 20 seconds.

SECONDARY OUTCOMES:
Self-identified countries of family origin up to grandparents | Within 10 minutes after consent to participate.
  The participant will report the countries which make up the participant's ancestral background, up to the country of origin of the grandparents.
A genotyped/imputed dataset of 8 million genetic variants aggregated using SHAPEIT (v2), IMPUTE2 (v2.3.2), Phase 3 1000 Genomes Project reference panel, SNP2HLA (v1.0.2), and the Type 1 Diabetes Genetics Consortium reference panel. | Saliva sample collected immediately after apnea, within 10min of propofol infusion start. Genomic analysis will be performed post-hoc.
  Extensive genome-wide genotyping to determine genetic variants of the pathways involved in propofol biotransformation. The array captures both common and rare variation collected from large-scale sequencing projects.

CONTACTS AND LOCATIONS:
Overall Officials: Simon Whyte, MBBS, FRCA, Principal Investigator — BC Children's Hospital, Department of Anesthesia
Locations (1):
- BC Children's Hospital - Department of Anesthesia, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Moxham L, Golam A, West NC, Gorges M, Whyte SD. Pharmacodynamic Safety Endpoints for Propofol Anesthesia in Children by Age and Sex: A Multicohort Observational Study. Paediatr Anaesth. 2025 Dec;35(12):1071-1079. doi: 10.1111/pan.70031. Epub 2025 Aug 11. PMID 40788031
- See also: Pediatric Anesthesia Research Team website — http://bcchr.ca/PART